CLINICAL TRIAL: NCT04674722
Title: Technetium-99m/Rhenium-188 Labeled Anti-HER2 Single Domain Antibody (99mTc/188Re-NM-02) for HER2 Expression Detection and Radionuclide Therapy in Breast Cancer
Brief Title: HER2 Expression Detection and Radionuclide Therapy in Breast Cancer Using 99mTc/188Re Labeled Single Domain Antibody
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: NanoMab Technology (UK) Limited (Industry)
Responsible Party: Principal Investigator, Zhao Jin Hua, MD, Director of Department of Nuclear Medicine, Principal Investigator, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020[84]
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Radiotoxicity
Keywords: HER2; single domain antibody; SPECT/CT imaging; Radionuclide therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of 99mTc-NM-02 (Experimental): All breast cancer patients recruited to the study will be administered 3-12 MBq/kg of 99mTc-NM-02 (99mTc labeled anti-HER2 sdAb) in a single dose injection.
  Interventions: Drug: Injection of 99mTc-NM-02
- Injection of 188Re-NM-02 (Experimental): Ten breast cancer patients recruited to the study will be administered 66 MBq/kg of 188Re-NM-02 (188Re labeled anti-HER2 sdAb) in a single dose injection.
  Interventions: Drug: Injection of 188Re-NM-02

INTERVENTIONS:
Drug: Injection of 99mTc-NM-02 — A Patient will be injected with microdose (<100ug) of 99mTc-NM-02 radiotracer
  Other Names: anti-HER2 SPECT/CT radiotracer
  Arms: Injection of 99mTc-NM-02
Drug: Injection of 188Re-NM-02 — A Patient will be injected with microdose (<100ug) of 188Re-NM-02 radionuclide therapy
  Other Names: anti-HER2 radionuclide therapy
  Arms: Injection of 188Re-NM-02

SUMMARY:
To evaluate the safety, dosimetry and efficacy of 99mTc/188Re labeled anti-HER2-single domain antibody (Product Code Name: 99mTc-NM-02 and 188Re-NM-02) SPECT/CT imaging of HER2 expression and radionuclide therapy in Breast Cancer. The SPECT/CT results will compare with the existing gold standard " HER2 expression detection" by biopsy tissue immunohistochemistry (IHC) and/or Fluorescence in Situ Hybridization (FISH) method, and 18F-FDG PET/CT imaging. It also to establish a new theranostic method for non-invasive HER2 expression detection and radionuclide therapy in breast cancer using 99mTc/188Re labeled anti-HER2 single domain antibody.

DETAILED DESCRIPTION:
Anti-HER2 single domain antibody will be labeled with 99mTc and 188Re to prepare 99mTc-NM-02 and 188Re-NM-02, respectively. 99mTc-NM-02 is used as a diagnostic agent for SPECT/CT imaging of HER2 expression, and 188Re-NM-02 is used as a therapeutic drug for radionuclide therapy of HER2-postive Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female, age 18 years or older
2. Prior diagnosis of breast cancer
3. Willing to participate in this study and given written informed consent
4. AST, ALT, BUN, Cr not more than double the normal values
5. Subjects of childbearing potential must be willing to undergo a pregnancy test prior to enrolment

Patients will only be included in the 188Re-NM-02 study if they meet the following supplementary criterial: HER2 postive, progression or recurrence after standard treatment, including surgery, chemotherapy, radiotherapy and targeted therapy.

Exclusion Criteria:

1. Pregnancy (subjects with a positive pregnancy test at baseline screening period or who are planning to become pregnant during the study period)
2. Breastfeeding (subjects in lactation)
3. No biopsy tissue sample can be provided for HER2 expression detection
4. Subjects with pacemakers
5. Hepatitis B virus infection (including carriers) at screening, ie hepatitis B surface antigen (HBsAg) positive, or hepatitis C antibody (anti-HCV) positive, or acquired immunodeficiency disease (HIV) infected, or serum syphilis positive person
6. Abnormal liver function during baseline screening period : AST or ALT> 2 times the upper limit of normal value (ULN), if the marginal increase of a single index is judged as having no clinical significance by the investigator, it can be retested during the screening period. Once, if ≤ 2 times ULN after retesting, consider enrolling).
7. Impaired renal function during screening: serum creatinine or urea nitrogen > 1.5 times ULN.
8. Within 4 months prior to the baseline screening period , myocardial infarction or other cardiac events requiring hospitalization (unstable angina, etc.), cerebrovascular accident, transient ischemic attack, acute congestive Heart failure or severe arrhythmia (ventricular arrhythmia, atrioventricular block above II)
9. Subjects with pulmonary embolism or deep vein thrombosis
10. Various infections that the investigators consider unsuitable for study, including but not limited to patients with various infections requiring further treatment, such as urinary tract infections, respiratory infections, and diabetic foot infections.
11. Patients with abnormal thyroid function during baseline screening period (including but not limited to active hyperthyroidism, hypothyroidism or Hashimoto's thyroiditis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Visual Assessment of HER2 expression in Breast cancer using 99mTc-NM-02 SPECT/CT Scan | 1 year
  Visual analysis will be carried out by 4 experienced nuclear medicine physicians to observe the uptake of 99m-Tc-NM-02 in breast malignant lesions. A 4-point system will be used to interpret the scans for abnormalities. It is categorised as such: score 0, no abnormal increased uptake; score 1, low increased uptake; score 2, moderate increased uptake; score 3, high increased uptake. The lesion will be considered positive for malignancy if the score is 2 or higher.
Semiquantitative Assessment of Breast and other Metastatic Lesions in 99mTc-NM-02 SPECT/CT Scan | 2 years
  Each subject will be administered 3-12 MBq/kg of 99mTc-NM-02 and the semiquantitative analysis of the region of interest (ROI) will be performed in breast and other metastatic lesions. Higher level of HER2 expression (Tumor proportion score, TPS), higher ROI in tumor.
  18F-FDG PET/CT, HER2 IHC and/or FISH used as comparators.
Safety of 99mTc-NM-02 through Adverse Event Monitoring | 2 years
  Subjects will be observed for safety after administration of 99mTc-NM-02, and will do follow up at 7 days p.i. Subjects will do blood test to observe for abnormalities in clinical parameters and compare to baseline results.
Changes of 99mTc-NM-02 uptake | 2 years
  The changes of tumor volume and maximum standard uptake value (SUVmax) will be recorded in primary and metastatic lesions
Safety of 188Re-NM-02 through Adverse Event Monitoring | 2 years
  Subjects will be observed for safety after administration of 188Re-NM-02, and will do follow up at 28 days p.i. Subjects will be contacted by investigator by phone and asked several questions related to subject's health after 188Re-NM-02 injection and concomitant drugs.

SECONDARY OUTCOMES:
Therapeutic evaluation of HER2 overexpressed Breast Cancer using 188Re-NM-02 | 3 years
  Ten patients will be administered 66 MBq/kg of 188Re-NM-02, and the changes of tumor volume and maximum standard uptake value (SUVmax) will be recorded in breast and other metastatic lesions to analyze treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Zhao, PhD, Principal Investigator — Department of Nuclear Medicine, Shanghai General Hospital
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Harbeck N, Gnant M. Breast cancer. Lancet. 2017 Mar 18;389(10074):1134-1150. doi: 10.1016/S0140-6736(16)31891-8. Epub 2016 Nov 17. PMID 27865536
- [Background] Keyaerts M, Xavier C, Heemskerk J, Devoogdt N, Everaert H, Ackaert C, Vanhoeij M, Duhoux FP, Gevaert T, Simon P, Schallier D, Fontaine C, Vaneycken I, Vanhove C, De Greve J, Lamote J, Caveliers V, Lahoutte T. Phase I Study of 68Ga-HER2-Nanobody for PET/CT Assessment of HER2 Expression in Breast Carcinoma. J Nucl Med. 2016 Jan;57(1):27-33. doi: 10.2967/jnumed.115.162024. Epub 2015 Oct 8. PMID 26449837
- [Background] Baum RP, Prasad V, Muller D, Schuchardt C, Orlova A, Wennborg A, Tolmachev V, Feldwisch J. Molecular imaging of HER2-expressing malignant tumors in breast cancer patients using synthetic 111In- or 68Ga-labeled affibody molecules. J Nucl Med. 2010 Jun;51(6):892-7. doi: 10.2967/jnumed.109.073239. Epub 2010 May 19. PMID 20484419
- [Derived] Zhao L, Xing Y, Liu C, Ma S, Huang W, Cheng Z, Zhao J. Detection of HER2 expression using 99mTc-NM-02 nanobody in patients with breast cancer: a non-randomized, non-blinded clinical trial. Breast Cancer Res. 2024 Mar 8;26(1):40. doi: 10.1186/s13058-024-01803-y. PMID 38459598